CLINICAL TRIAL: NCT01793454
Title: Comparing the Effect of Hyperoxic and Conventional Fraction of Inspired Oxygen on Oxidative Stress During Abdominal Surgery.
Brief Title: Hyperoxic Oxidative Stress During Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Assoc.Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36048
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Response to Hyperoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 40% oxygen (Active Comparator): Patients in this group will be ventilated with fraction of inspired oxygen 40% during the surgery.
  Interventions: Other: Fraction of inspired oxygen 40%
- 80% oxygen (Active Comparator): Patients in this group will be ventilated with a fraction of inspired oxygen 80% during the surgery.
  Interventions: Other: Fraction of inspired oxygen 80%

INTERVENTIONS:
Other: Fraction of inspired oxygen 40%
  Arms: 40% oxygen
Other: Fraction of inspired oxygen 80%
  Arms: 80% oxygen

SUMMARY:
Our aim is to compare the effects of 80% and 40% Fraction of inspired oxygen on oxidative stress, antioxidant response (in plasma and bronchoalveolar lavage), extubation quality, preanesthetic and postanesthetic expiration tidal volumes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal surgery, between 20-60 years old, with American Society of Anesthesiology score I or II

Exclusion Criteria:

* Patients with Chronic Obstructive Pulmonary Disease, Diabetes Mellitus, muscle-bone diseases, inflammatory bowel diseases and patients with malnutrition.

Patients will be recruited through general surgery service of our hospital

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
oxidant and antioxidant response | 4 hours
  As primary outcome, the effects of different inspired oxygen fractions on oxidative stress and anti-oxidant response in plasma and bronchoalveolar lavage after intubation and prior to extubation will be evaluated

SECONDARY OUTCOMES:
Hemodynamics | 4 hours
  The secondary outcome was evaluating the effects of different inspired oxygen fractions on hemodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Yalim Dikmen, Prof., Study Director — Cerrahpasa Medical Faculty Chairman of Intensive Care Department
Locations (1):
- Cerrahpasa Medical Faculty Anesthesiology and Reanimation Department, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Koksal GM, Sayilgan C, Aydin S, Uzun H, Oz H. The effects of sevoflurane and desflurane on lipid peroxidation during laparoscopic cholecystectomy. Eur J Anaesthesiol. 2004 Mar;21(3):217-20. doi: 10.1017/s0265021504003102. PMID 15055896